CLINICAL TRIAL: NCT02309697
Title: Neurodevelopmental Outcomes of Preterm and Term Children
Status: Terminated | Type: Observational
Why Stopped: Study goals rolled into a broader study
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: GCO 12-0332-0001
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Development
Keywords: Development; Assessments; Premature birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Full Term: Children born at full term on or after Jan 1, 2011
- PreTerm: Children born preterm on or after Jan 1, 2011

SUMMARY:
This study will utilize two validated tools for assessing child development and behavior, to investigate the outcomes for children born preterm compared with those born at full term. Two hundred children born or cared for during the neonatal period at Mount Sinai Hospital will be enrolled. Parents will be asked to complete a behavioral assessment questionnaire, and which will assess development in an examination administered by a trained occupational therapist at Mount Sinai Hospital.

DETAILED DESCRIPTION:
This research will be completed at Mount Sinai Hospital. All participants will be identified from Mount Sinai Hospital records of infants born at MSH and/or cared for in the Mount Sinai NICU on or after January 1, 2011, at full term or preterm. The study team will contact the parents of eligible potential participants by telephone to explain the study and ask if the parent will consent to their child's participation. If the parent agrees, we will make an appointment for the child to come to Mount Sinai for the evaluation using the Bayley-III. The parents will be mailed the study consent form, a fact sheet with information about the study, and the CBCL to complete before they bring their child to their appointment. Mount Sinai records from the birth hospitalization will be reviewed for the birth history and medical comorbidities. Mount Sinai medical records of the mother's obstetric care will also be accessed to obtain medical history from the pregnancy. If a participating child has received outpatient care at Mount Sinai, the investigators will access their record in Epic to obtain scores from previous developmental assessments and records of medical comorbidities. If they have not attended the Mount Sinai clinic, but have received outpatient care elsewhere, the parents will be asked to provide contact information for their pediatrician, and for permission to obtain their child's records.

ELIGIBILITY:
Inclusion Criteria:

* Born on or after January 1, 2011
* Admitted to the Mount Sinai Hospital for newborn care

Exclusion Criteria:

* Non-English speaking

Ages: 6 Months to 42 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 200 children born on or after January 1, 2011 at Mount Sinai or admitted to the Mount Sinai Hospital for newborn care.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2015-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Child Behavior Checklist (CBCL) | day 1
  The CBCL, completed by a primary caregiver, is a standardized assessment of behavioral problems categorized into externalizing or internalizing behaviors.

SECONDARY OUTCOMES:
Bayley Scales of Development III (BayleyIII) | day 1
  The Bayley Scales of Infant and Toddler Development, Third Edition (Bayley-III) is used to measure developmental and behavioral outcomes. The Bayley-III is a standardized assessment of cognitive, motor, and language development administered by a trained researcher. The Bayley-III also includes social and emotional development questionnaire that is completed by a primary caregiver.

CONTACTS AND LOCATIONS:
Overall Officials: Annemarie Stroustrup, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States